CLINICAL TRIAL: NCT00889915
Title: A Randomized Controlled Trial of Methylphenidate Transdermal System (Daytrana), Lisdexamfetamine Dimesylate (Vyvanse), OROS MPH (Concerta), and Mixed Amphetamine Salts Extended Release (Adderall XR) in Children and Adolescents With ADHD
Brief Title: Comparing the Effectiveness of New Versus Older Treatments for Attention Deficit Hyperactivity Disorder (The NOTA Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014075; P30MH066386-02 (NIH); DSIR CTM 4571; Pro00014075
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Methylphenidate; Amphetamine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Lisdexamfetamine Dimesylate; SLI381

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Participants will receive methylphenidate transdermal system.
  Interventions: Drug: Methylphenidate transdermal system
- 2 (Active Comparator): Participants will receive lisdexamfetamine dimesylate.
  Interventions: Drug: Lisdexamfetamine dimesylate
- 3 (Active Comparator): Participants will receive osmotic-release oral system methylphenidate (OROS MPH).
  Interventions: Drug: Osmotic-release oral system methylphenidate (OROS MPH)
- 4 (Active Comparator): Participants will receive mixed amphetamine salts extended release.
  Interventions: Drug: Mixed amphetamine salts extended release

INTERVENTIONS:
Drug: Methylphenidate transdermal system — Not specified in protocol; determined by local standard of care.
  Other Names: Daytrana
  Arms: 1
Drug: Lisdexamfetamine dimesylate — Not specified in protocol; determined by local standard of care.
  Other Names: Vyvanse
  Arms: 2
Drug: Osmotic-release oral system methylphenidate (OROS MPH) — Not specified in protocol; determined by local standard of care.
  Other Names: Concerta
  Arms: 3
Drug: Mixed amphetamine salts extended release — Not specified in protocol; determined by local standard of care.
  Other Names: Adderall XR
  Arms: 4

SUMMARY:
This study will determine whether two new psychostimulant medications are more effective, tolerable, and acceptable than two older medications for treating attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is characterized by impulsiveness, hyperactivity, and inattention. It is seen primarily in children and adolescents and is often treated with psychostimulant medications. Osmotic-release oral system (OROS) methylphenidate, brand name Concerta, and mixed amphetamine salts extended release, brand name Adderall XR, are psychostimulant medications that have shown both efficacy (that they can have therapeutic benefits) and effectiveness (that they typically have therapeutic benefits in practice). Two newer psychostimulant medications-lisdexamfetamine dimesylate, brand name Vyvanse, and methylphenidate transdermal system, brand name Daytrana-have shown efficacy but have not been tested for effectiveness, nor have they been tested head-to-head against the older psychostimulants. This study will test the effectiveness, tolerability (lack of side effects), and acceptability (ease of use for patients) of the two newer psychostimulant medications and compare them to each other and to the two older psychostimulants.

Participation in this study will last 6 weeks, although some treatments may continue past the end of the study. At enrollment, participants will undergo a series of baseline evaluations. These will include interviews and assessments of ADHD symptoms, concurrent psychiatric disorders, medical and psychiatric history, family history of mental illness, risk and protective factors, other treatments, treatment expectancy of both the youth and parent, and vital signs. In consultation with their doctors, participants will be allowed to exclude zero, one, or two of the study medications; if they choose to exclude both of the new ADHD medications, they will not able to participate in the study. Participants will then be randomly assigned to one of the treatments they choose to include. They will receive a prescription for the medication and instructions for how to use it from their doctors; the study protocol does not specify a particular treatment regimen. Participants will undergo a second set of evaluations after 6 weeks of treatment or before, if the treatment ends earlier. This will include interviews and assessments similar to those administered at baseline as well as evaluation of any medication side effects.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnostic criteria for ADHD combined, hyperactive/impulsive, or inattentive subtype
* Outpatient at study entry
* Speaks English
* Willing to be randomly assigned to one of the study treatment options as outlined in the protocol
* No known significant history of cardiovascular disorders, including pre-existing congenital heart disease, structural heart disease, known clinically significant electrocardiogram (ECG) abnormality, or other clinically significant cardiac disorder
* Willing to initiate study medication for ADHD within 7 days of the study baseline visit
* May be receiving stable treatment with other drug for a comorbid disorder, defined as no changes in dose or form of drug treatment for at least 2 weeks prior to the study enrollment visit
* May be receiving psychosocial interventions for ADHD or a comorbid disorder, defined as no changes in form of psychosocial treatment for at least 4 weeks prior to the study enrollment visit

Exclusion Criteria:

* Hypersensitivity to study medication
* Inpatient status at study entry
* Currently taking another medication for ADHD, including another psychostimulant, atomoxetine, or bupropion
* Receiving treatment with a tricyclic antidepressant at study enrollment, with the exception of low-dose imipramine for enuresis or amitriptyline for chronic pain
* Received treatment with a monoamine oxidase inhibitor (MAOI) within the past 30 days
* Psychostimulant drug dependence, bipolar disorder, or schizophrenia
* Presence of psychosis
* Severe mental retardation
* Autism or Asperger's syndrome
* Active suicidal ideation
* Unable or unwilling to comply with the protocol
* Demonstrates a lack of benefit from, an intolerance to, or contraindication to psychostimulant medicine
* Presence of other clinically significant medical conditions, including hyperthyroidism, epilepsy or other seizure disorder, any condition for which an increase in blood pressure or heart rate would be problematic, glaucoma or other significant eye disease for which a psychostimulant would be problematic, or pre-existing gastrointestinal obstruction with gastrointestinal narrowing
* Pregnant or positive result of pregnancy test

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 228 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S. March, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Child and Adolescent Psychiatry Trials Network (CAPTN), Durham, North Carolina, United States

REFERENCES:
- See also: Click here for the Duke Clinical Research Institute Web site — http://dcri.org/
- See also: Click here for the American Academy of Child and Adolescent Psychiatry Web site — http://www.aacap.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was April to October 2009. Recruitment occurred at Child and Adolescent Psychiatry clinics in the USA.
Groups:
- Daytrana (Methylphenidate Transdermal System: Participants will receive methylphenidate transdermal system.
  Methylphenidate transdermal system : Not specified in protocol; determined by local standard of care.
- Vyvanse (Lisdexamfetamine Dimesylate): Participants will receive lisdexamfetamine dimesylate.
  Lisdexamfetamine dimesylate : Not specified in protocol; determined by local standard of care.
- Concerta (Osmotic-release Oral System Methylphenidate): Participants will receive osmotic-release oral system methylphenidate (OROS MPH).
  Osmotic-release oral system methylphenidate (OROS MPH) : Not specified in protocol; determined by local standard of care.
- Adderall (Mixed Amphetamine Salts Extended Release): Participants will receive mixed amphetamine salts extended release.
  Mixed amphetamine salts extended release : Not specified in protocol; determined by local standard of care.
Period: Overall Study
Arm/Group | Daytrana (Methylphenidate Transdermal System | Vyvanse (Lisdexamfetamine Dimesylate) | Concerta (Osmotic-release Oral System Methylphenidate) | Adderall (Mixed Amphetamine Salts Extended Release)
Started | 37 | 76 | 67 | 48
Completed | 35 | 71 | 54 | 40
Not Completed | 2 | 5 | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Daytrana (Methylphenidate Transdermal System: Participants will receive methylphenidate transdermal system. Although not specified by protocol, rather determined by local standard of care, the typical doses and strategies are as follows:
  Dose form as 10, 15, 20, 30 mg patches. Typical starting dose is 10 mg patch every day then titrate up by patch strength.
  The FDA maximum dose per day is 30 mg and the off label maximum dose per day is 40 mg.
  The patch should be applied to the hip area, avoiding the waistline and the patch application should be alternated between hips.
- Vyvanse (Lisdexamfetamine Dimesylate): Participants will receive lisdexamfetamine dimesylate.
  Although not specified by protocol, rather determined by local standard of care, the typical doses and strategies are as follows:
  Dose form is 20, 30, 40, 50, 60, 70 mg ivory body/ivory cap. The typical starting dose is 30 mg every day in the morning; dosage may be adjusted in increments of 10 mg or 20 mg at approximately weekly intervals.
  The FDA maximum dose per day is 70 mg. Afternoon doses should be avoided because of the potential for insomnia. Vyvanse may be taken with or without food. Vyvanse capsules may be taken whole, or the capsule may be opened and the entire contents dissolved in a glass of water. The solution should be consumed immediately and should not be stored. The dose of a single capsule should not be divided.
- Concerta (Osmotic-release Oral System Methylphenidate): Participants will receive osmotic-release oral system methylphenidate (OROS MPH).
  Although not specified by protocol, rather determined by local standard of care, the typical doses and strategies are as follows:
  Dose form is 18, 27, 36, 54 mg capsules. The typical starting dose is 18 mg every morning. The FDA maximum dose per day is 54 mg in children or 72 mg in adolescents. The off label maximum dose is 108 mg. Longer acting stimulants offer greater convenience, confidentiality, and compliance with single daily dosing, but may have greater problematic effects on evening appetite and sleep. Its nonabsorbable tablet shell may appear in the stool.
  Osmotic-release oral system methylphenidate (OROS MPH) : Not specified in protocol; determined by local standard of care.
- Adderall (Mixed Amphetamine Salts Extended Release): Participants will receive mixed amphetamine salts extended release.
  Although not specified by protocol, rather determined by local standard of care, the typical doses and strategies are as follows:
  The dose form for is 5, 10, 15, 20, 25, 30 mg capsules. The typical starting dose for children greater than or equal to 6 years of age is 10 mg every day.
  The FDA maximum dose per day is 30 mg if weight is greater than 50 kilograms. The off label maximum dose per day is 60 mg. The capsule may be opened and sprinkled on soft foods.
- Total: Total of all reporting groups
Arm/Group | Daytrana (Methylphenidate Transdermal System | Vyvanse (Lisdexamfetamine Dimesylate) | Concerta (Osmotic-release Oral System Methylphenidate) | Adderall (Mixed Amphetamine Salts Extended Release) | Total
Number analyzed (Participants) | 37 | 76 | 67 | 48 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 76 | 67 | 48 | 228
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.3 (3.2) | 10.6 (3.1) | 10.0 (3.2) | 10.4 (3.0) | 10.3 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 21 | 25 | 16 | 72
  Male | 27 | 55 | 42 | 32 | 156
Region of Enrollment [Number; unit: participants]
  United States | 37 | 76 | 67 | 48 | 228

OUTCOME MEASURES:

1. Primary Outcome: Dichotomized Clinical Global Impression-Effectiveness (CGI-E) Scale
Description: The CGI-E is the value at which the participant's Therapeutic Benefit and Adverse Impact to the study drug intersect. This number is determined by combining each participant's scores for the degree of Therapeutic Benefit versus the degree to which problems with Tolerability and/or Acceptability adversely impact the subject. Participants are then determined to be Responders or Non-responders to the study medication. For example, a subject who is very much improved (CGI-I=1) or much improved (CGI-I=2) therapeutically and whose adverse impact rating is none (score 1,5) or mild (score 2,6) will be categorized as a Responder. All others whose adverse impact rating is moderate (score 3,7,11,15)or outweighs therapeutic effect (score 4,8,12,16) will be categorized as Non-responders to study medication. The CGI scores are totaled for each participant and a mean score is calculated. A median total score was calculated for each treatment group.
Time Frame: Measured at each participant's last visit, which can occur at or before Week 6
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Daytrana (Methylphenidate Transdermal System | Vyvanse (Lisdexamfetamine Dimesylate) | Concerta (Osmotic-release Oral System Methylphenidate) | Adderall (Mixed Amphetamine Salts Extended Release)
Number analyzed (Participants) | 35 | 71 | 54 | 40
Units on a scale | 7.0 (16.0) [1.0 to 16.0] | 5.0 (16.0) [1.0 to 16.0] | 6.0 (16.0) [1.0 to 16.0] | 6.0 (16.0) [1.0 to 16.0]

2. Secondary Outcome: Clinical Global Impressions-Improvement (CGI-I) Scale
Description: The CGI-I score at the subject's last study visit at or before Week 6, is one of the 3 secondary endpoints that contribute to the primary endpoint (CGI-E). The CGI-I scale will be used to rate improvement in the subject's condition (benefits) since baseline using the following 7-point scale: 1=very much improved, 2=much improved, 3=minimally improved, 4=not changed, 5=minimally worse, 6=much worse; 7=very much worse.
Time Frame: Measured at each participant's last visit, which can occur at or before Week 6
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Daytrana (Methylphenidate Transdermal System | Vyvanse (Lisdexamfetamine Dimesylate) | Concerta (Osmotic-release Oral System Methylphenidate) | Adderall (Mixed Amphetamine Salts Extended Release)
Number analyzed (Participants) | 35 | 71 | 54 | 40
Units on a scale | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 5.0]

3. Secondary Outcome: Clinical Global Improvements-Acceptability (CGI-A) Scale
Description: The CGI-A score at the subject's last study visit at or before Week 6 is one of the 3 secondary endpoints that contribute to the primary endpoint (CGI-E). The CGI-A will be used to assess the acceptability of the study medication with respect to the subject's experience with the formulation of medication. The 7-point rating for the CGI-A will be: 1=very high acceptability, 2=high acceptability, 3=above average acceptability, 4=average acceptability, 5=low acceptability, 6=very low acceptability, 7=extremely low acceptability
Time Frame: Measured at each participant's last visit, which can occur at or before Week 6
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Daytrana (Methylphenidate Transdermal System | Vyvanse (Lisdexamfetamine Dimesylate) | Concerta (Osmotic-release Oral System Methylphenidate) | Adderall (Mixed Amphetamine Salts Extended Release)
Number analyzed (Participants) | 35 | 71 | 54 | 40
Units on a scale | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline through the participant's last visit. The participant's last visit can can occur at or before 6 weeks after study medication was started.
Arm/Group | Daytrana (Methylphenidate Transdermal System | Vyvanse (Lisdexamfetamine Dimesylate) | Concerta (Osmotic-release Oral System Methylphenidate) | Adderall (Mixed Amphetamine Salts Extended Release)
Serious Adverse Events (participants affected / at risk) | 2/33 | 0/67 | 1/53 | 0/39
Other Adverse Events (participants affected / at risk) | 16/33 | 33/67 | 18/53 | 15/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Daytrana (Methylphenidate Transdermal System (N=33) | Vyvanse (Lisdexamfetamine Dimesylate) (N=67) | Concerta (Osmotic-release Oral System Methylphenidate) (N=53) | Adderall (Mixed Amphetamine Salts Extended Release) (N=39)
Tachycardia / arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Assaultive/Aggressive behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0/52 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daytrana (Methylphenidate Transdermal System (N=33) | Vyvanse (Lisdexamfetamine Dimesylate) (N=67) | Concerta (Osmotic-release Oral System Methylphenidate) (N=53) | Adderall (Mixed Amphetamine Salts Extended Release) (N=39)
Irritability (Psychiatric disorders) | 1 (9) | 5 (9) | 1 (9) | 2 (9)
Insomnia (Psychiatric disorders) | 5 (18) | 6 (18) | 5 (18) | 2 (18)
Angry or hostile mood (Psychiatric disorders) | 1 (9) | 3 (9) | 2 (9) | 3 (9)
Weight loss (General disorders) | 2 (10) | 3 (10) | 3 (10) | 2 (10)
Decreased appetite (General disorders) | 5 (25) | 11 (25) | 4 (25) | 5 (25)
Emotional lability (Psychiatric disorders) | 2 (9) | 4 (9) | 2 (9) | 1 (9)
Tics (Nervous system disorders) | 2 (2) | 1 (2) | 1 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No